CLINICAL TRIAL: NCT05439824
Title: A Randomized, Observer-blinded, Placebo-Controlled Phase 2 Clinical Study to Evaluate the Immunogenicity and Safety of a SARS-CoV-2 mRNA Vaccine (SYS6006) in Healthy Participants Aged 18 Years or More
Brief Title: A Study of SARS-CoV-2 mRNA Vaccine (SYS6006) in Chinese Healthy Participants Aged 18 Years or More
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SYS6006-003
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — SYS6006 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20 μg dose of SYS6006 (Aged 18~59 years or 60 years or more) (Experimental): 20μg dose of SYS6006 vaccine IM, on day 0 and day 21.
  Interventions: Biological: SYS6006 20 μg
- 30 μg dose of SYS6006 (Aged 18~59 years or 60 years or more) (Experimental): 30 μg dose of SYS6006 vaccine IM, on day 0 and day 21.
  Interventions: Biological: SYS6006 30 μg
- Placebo(Aged 18~59 years or 60 years or more) (Placebo Comparator): placebo IM, on day 0 and day 21 .
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SYS6006 20 μg — SARS-CoV-2 mRNA Vaccine
  Arms: 20 μg dose of SYS6006 (Aged 18~59 years or 60 years or more)
Biological: SYS6006 30 μg — SARS-CoV-2 mRNA Vaccine
  Arms: 30 μg dose of SYS6006 (Aged 18~59 years or 60 years or more)
Biological: Placebo — Placebo
  Arms: Placebo(Aged 18~59 years or 60 years or more)

SUMMARY:
This is a phase 2, randomized, observer-blinded, placebo-controlled clinical study to evaluate the immunogenicity and safety of SARS-CoV-2 mRNA Vaccine (SYS6006）in healthy participants aged 18 or more.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of the first dose of vaccine: 18 and above;
2. Axillary body temperature is less than 37.3 degree centigrade on the day of enrollment;
3. Based on the medical history, physical examination and laboratory examination results, the investigator clinically determined the qualified person.
4. Has independent judgment, and participate voluntarily and sign an informed consent form.

Exclusion Criteria:

* Those who meet any of the following criteria must be excluded from this study:

  1. Has a history of SARS or SARS-CoV-2 infection, or close contact with SARS-CoV-2 infected person( nucleic acid test positive), or living abroad within 30 days before screening;
  2. Positive for SARS-CoV-2 antibody test;
  3. History of allergy to paracetamol or vaccination (such as acute allergic reaction, urticaria, dyspnea, angioedema, or abdominal pain);
  4. Has a history of vaccination with SARS-CoV-2 vaccine, or vaccination with other inactivated or recombinant vaccine within 7 days or received live attenuated vaccine within 14 days before the first dose;
  5. Has a medical or family history of epilepsy or convulsion, neurological disorders, mental disorders, etc.;
  6. Is contraindications for intramuscular injection, such as diagnosed thrombocytopenia, any coagulation disorder or receiving anticoagulant treatment, etc.;
  7. Has known or suspected serious disorders judged by the Investigator, including but not limited to respiratory disorders (pulmonary failure, etc.), liver and kidney disorders, cardiovascular disorders (cardiac failure, severe hypertension, etc.), malignant tumors, infections or allergic skin disorders, HIV infection, or in the acute infection or chronic disease activity period (within 3 days before vaccination);
  8. Has chronic diseases (such as Down syndrome, sickle cell anemia, neurological disorders and Guillain-Barre syndrome, excluding chronic diseases such as controlled stable diabetes mellitus/hypertension/hyperlipidemia) that are not suitable for this study at the discretion of the Investigator;
  9. Has known immunological impairment or immunodeficiency diagnosed by hospital before enrollment, or functional asplenia or splenectomy caused by any condition;
  10. For women of childbearing potential: positive pregnancy test before the enrollment, being in pregnant, breastfeeding, or have a pregnancy plan within 1 year; men: whose spouses is of childbearing potential and has a pregnancy plan within 1 year;
  11. Is participating or plan to participate in other clinical studies during the study;
  12. Has received immune enhancement or immunosuppressive therapy within 3 months (continuous oral or instillation for more than 14 days); or received treatment with whole blood, plasma and immunoglobulin within 1 month;
  13. Is unlikely to adhere to the study procedures or keep appointments at the discretion of the investigators;or has other conditions that are not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-06-28 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT), geometric mean increase (GMI) and seroconversion rate (SCR) of serum anti-SARS-CoV-2 neutralizing antibody and IgG antibody | 14 days after the second dose
Adverse events (AEs), including solicited AEs and unsolicited AEs | From the first dose through 30 days following the second dose
AEs associated with the study intervention | From the first dose through 30 days following the second dose

SECONDARY OUTCOMES:
Serious adverse events (SAEs) | from the first dose through 12 months after the second dose.
Adverse events of special interest (AESIs) | rom the first dose through 12 months after the second dose.
Laboratory test related adverse events | 4 days following each dose.
Geometric Mean Titer(GMT), Geometric Mean Fold Increase (GMI) and Seroconversion Rate (SCR) of serum anti-SARS-CoV-2 neutralizing antibody and IgG antibody | from the first dose through 21 days
GMT, GMI and SCR of serum anti-SARS-CoV-2 neutralizing antibody and IgG antibody | 30, 90, 180 and 360 days after the second dose.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliang Zhao, Principal Investigator — Center For Disease Control and Prevention, Hebei Province; Jingxin Li, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention; Xiang Lu, Principal Investigator — Nanjing Medical University
Locations (2):
- China (2):
  - Hebei Provincial Center For Disease Control and Prevention, Shijiazhuang, Hebei
  - Sir Run Run Hosipital Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No